CLINICAL TRIAL: NCT00005525
Title: Sleep Apnea in Elderly Male Twins
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5053; R01HL059659 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2005-03

CONDITIONS: Lung Diseases; Sleep Apnea Syndromes; Obesity
MeSH Terms: conditions — Lung Diseases; Sleep Apnea Syndromes; Obesity

SUMMARY:
To conduct a genetic analysis of anatomic risk factors for sleep apnea in a well-characterized United States population-based registry of elderly male twins who have been successfully followed for the past 30 years.

DETAILED DESCRIPTION:
BACKGROUND:

The contribution of genetic factors to sleep disorders has been demonstrated in twin and family studies, and further understanding of the genetic underpinning of sleep disorders is considered an important area of research. Many of the suggested risk factors for sleep apnea (e.g.,craniofacial morphology, obesity) have genetic determinants. However, a formal genetic analysis of these anatomical risk factors with sleep-recorded physiological measurements has not so far been conducted.

DESIGN NARRATIVE:

The investigators recruited a subsample of pairs from the NAS-NRC World War II Twin Registry in which at least one of the twin brothers reported sleep apnea symptoms and a subsample of control pairs in which both twins reported no symptoms. They monitoring the subgroup of twin pairs with overnight sleep recording. They also collected anthropometric measurements of weight, height, neck circumference, and craniofacial morphology and blood samples for determination of zygosity and DNA extraction for future molecular studies.

The twin design is most powerful for estimating the genetic and/or environmental overlap between physiological measurements such as sleep-recorded disordered breathing, obesity, and craniofacial morphology. The investigators chose to focus on an elderly male twin sample for which a wealth of data relevant to this study had been previously collected. Twin pair concordance or discordance for monitored sleep-disordered breathing allowed the full characterization of genetic/familial and individual environmental factors associated with the expression and severity of this condition.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-08; Study Completion 2002-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dorit Carmelli — SRI International

REFERENCES:
- [Background] Carmelli D, Bliwise DL, Swan GE, Reed T. A genetic analysis of the Epworth Sleepiness Scale in 1560 World War II male veteran twins in the NAS-NRC Twin Registry. J Sleep Res. 2001 Mar;10(1):53-8. doi: 10.1046/j.1365-2869.2001.00241.x. PMID 11285055
- [Background] Carmelli D, Bliwise DL, Swan GE, Reed T. Genetic factors in self-reported snoring and excessive daytime sleepiness: a twin study. Am J Respir Crit Care Med. 2001 Sep 15;164(6):949-52. doi: 10.1164/ajrccm.164.6.2012001. PMID 11587976
- [Background] Carmelli D, Colrain IM, Swan GE, Bliwise DL. Genetic and environmental influences in sleep-disordered breathing in older male twins. Sleep. 2004 Aug 1;27(5):917-22. doi: 10.1093/sleep/27.5.917. PMID 15453550